CLINICAL TRIAL: NCT06837909
Title: Transversus Abdominis Plane Block Versus Wound Infiltration for Pulmonary Function Preservation Following Laparoscopic Living Donor Nephrectomy (The TAPWIN Trial): A Double-Blind Randomized Controlled Trial
Brief Title: Transversus Abdominis Plane Block Versus Wound Infiltration for Pulmonary Function Preservation Following Laparoscopic Living Donor Nephrectomy
Acronym: TAPWIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, karam azem, Attending Anesthesiologist, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0131-25-RMC
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Operating room staff (anesthesiologists and surgeons) are unblinded due to the nature of the interventions. Patients, the physician measuring peak expiratory flow, PACU staff, and transplantation surgical ward nursing staff are blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP Block Group (Experimental): After anesthesia induction and before surgical incision, the anesthesiologist will perform an ultrasound-guided (Venue GO, GE Healthcare, USA) single-shot TAP block in the triangle of Petit with 20 mL 0.25% bupivacaine and 2.5 µg mL-1 of epinephrine on each side.
  Interventions: Procedure: Transversus abdominis plane (TAP) block
- Wound Infiltration Group (Active Comparator): Following surgery conclusion and before awakening from anesthesia, the surgeons will inject 40 mL of 0.25% bupivacaine and 2.5 µg mL-1 of epinephrine at the wound sites.
  Interventions: Procedure: Wound infiltration

INTERVENTIONS:
Procedure: Transversus abdominis plane (TAP) block — A regional anesthesia technique in which a local anesthetic is injected into the transversus abdominis plane under ultrasound guidance to provide postoperative analgesia.
  Arms: TAP Block Group
Procedure: Wound infiltration — A local anesthetic technique where bupivacaine with epinephrine is injected directly into the surgical wound sites to provide postoperative analgesia.
  Arms: Wound Infiltration Group

SUMMARY:
This study compares two pain control techniques in patients undergoing laparoscopic kidney donation surgery: transversus abdominis plane (TAP) block versus wound infiltration with local anesthetic.

Postoperative pain can impair breathing by causing patients to take shallow breaths to avoid discomfort. This study will evaluate which technique better preserves lung function, specifically peak expiratory flow (PEF), after surgery.

Eighty patients will be randomly assigned to receive either a TAP block (injection of local anesthetic into the abdominal wall muscles before surgery) or wound infiltration (injection of local anesthetic at the incision sites at the end of surgery). Both patients and the staff measuring outcomes will be blinded to group assignment.

The primary outcome is the percentage change in PEF from before surgery to discharge from the recovery room. Secondary outcomes include pain scores, opioid use, breathing complications, and length of hospital stay.

DETAILED DESCRIPTION:
Laparoscopic living donor nephrectomy (LLDN) is the gold-standard approach for kidney donation, offering reduced pain, shorter hospital stays, and faster recovery compared to open surgery. However, postoperative pain remains a concern, particularly because acute pain leads to protective "splinting" breathing patterns - shallow, rapid breaths that limit abdominal wall movement. This restricted breathing reduces thoracic expansion, inhibits deep inspiration, and impairs effective coughing, increasing the risk of pulmonary complications.

Among regional analgesic techniques, TAP block and wound infiltration have emerged as promising options for LLDN due to their simplicity and effectiveness. TAP block involves ultrasound-guided injection of local anesthetic between the internal oblique and transversus abdominis muscles, providing analgesia to the anterolateral abdominal wall. Wound infiltration directly targets the surgical incision sites. While both techniques reduce postoperative pain and opioid consumption, their comparative effectiveness in preserving pulmonary function remains unclear.

This double-blind randomized controlled trial will compare the effects of TAP block versus wound infiltration on peak expiratory flow (PEF) preservation following LLDN. All patients will receive standardized general anesthesia and multimodal analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo elective LLDN.
* Age above 18 years.
* Body Mass Index (BMI) above 20 and below 40 kg m-2.
* Eligible to sign informed consent.

Exclusion Criteria:

* Open or hand-assisted surgery.
* Known cardiac or pulmonary disease.
* Preoperative chronic pain (i.e., fibromyalgia, chronic neuropathic pain).
* Contraindication for regional analgesia (i.e., known allergy to LA, skin lesions in the injection site).
* Known allergy to one or more of the components of multimodal analgesia (i.e., opioids, paracetamol, tramadol, dipyrone).
* Preexisting severe pulmonary disease (i.e., an obstructive lung disease with a forced expiratory volume in the first second [FEV1] below 49%, restrictive lung disease with a forced vital capacity [FVC] below 49%, pulmonary hypertension).

Discontinuing criteria:

Participants will be excluded from the analysis if they:

* Experience intraoperative bleeding requiring transfusion of more than three units of blood products.
* Experience hemodynamic instability requiring postoperative vasopressor or inotropic support.
* Require conversion to open surgery.
* Require mechanical ventilation after being transferred from the OR to the PACU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Peak Expiratory Flow (PEF) | Baseline (Preoperative) and PACU Discharge (Within 2-3 hours post-surgery)
  Percentage change in PEF (measured in liters per second) between preoperative baseline and post-anesthesia care unit discharge.

SECONDARY OUTCOMES:
Pain scores | Within 48 hours postoperatively
  Pain intensity measured using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate worse outcome.
Opioid Consumption | Within 48 hours postoperatively
  Opioid consumption, measured in morphine milligram equivalence (MME)
Incidence of postoperative pulmonary complications | From the day of surgery until hospital discharge (typically within 3-5 days postoperatively)
  Based on the European perioperative clinical outcome (EPCO) criteria.
Length of post-anesthesia care unit (PACU) stay | Typically within 6 hours postoperatively
  The total time (in hours) a patient remains in the PACU
Length of Hospital Stay | From the day of surgery until hospital discharge (typically within 3-5 days postoperatively)
  The total length of hospital stay (in days) from surgery until hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel